CLINICAL TRIAL: NCT03180125
Title: Use of Hyaluronic Acid Injection in Treatment of Idiopathic Carpal Tunnel Syndrome Versus Corticosteroid Injection Sonographically Guided
Brief Title: Hyaluronic Acid Hydro-dissection Use in Idiopathic Carpal Tunnel Syndrome Guided by Ultrasonic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyaluronic injection
Record Dates: First submitted 2016-07-11; First posted 2017-06-08 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: hydrodissection; sodium hyaluorinate
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Hyaluronic Acid; Ultrasonography; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- sodium hyaluorinate ultrasound guided (Experimental): median nerve hydro-dissection using 1% lidocain followed by low molecular weight sodium hyaluronate (Hyalgan) injection ultrasonographically guided
  Interventions: Drug: Sodium Hyaluronate; Device: ultrasound; Drug: Sodium Hyaluronate and 1% lidocain
- corticosteroid with ultrasound guided (Placebo Comparator): median nerve hydro-dissection using 1% lidocain followed by injection of corticosteroid Ultrasonographically guided
  Interventions: Device: ultrasound; Drug: Sodium Hyaluronate and 1% lidocain; Drug: Corticosteroid and 1%lidocain

INTERVENTIONS:
Drug: Sodium Hyaluronate — median nerve in CTS hydro-dissection using 1% lidocain followed by injection of Sodium hyaluronate guided by ultrasound
  Other Names: hyalgan
  Arms: sodium hyaluorinate ultrasound guided
Device: ultrasound — ultrasound guided injection
Drug: Sodium Hyaluronate and 1% lidocain — injection in the carpal tunnel
Drug: Corticosteroid and 1%lidocain — injection in the carpal tunnel
  Arms: corticosteroid with ultrasound guided

SUMMARY:
carpal tunnel syndrome (CTS) is the most common compression syndrome in the upper extremities, CTS is characterized by typical anatomic changes, the most probable swelling of the median nerve in the proximal part of the CT.

Local infiltration of corticosteroids easily leads to atrophy of the median nerve, subcutaneous fat, and systematic complications, surgical treatment decision is always taken by the patient who sometimes wants to delay or avoid the surgery because of psychological or medical concerns, It would be interesting if low molecular weight sodium hyaluorinate injection is used as an alternative conservative treatment of CTS. This study aims to investigate if, and to what extent, hydro-dissection using 1% lidocain followed by injection of Sodium hyaluronate versus 1% lidocain followed by injection of 40 mg of triamcinolone acetonide, under ultrasound guidance.

DETAILED DESCRIPTION:
60 CT patients, blindly divided into two groups. Both will underwent median nerve hydro-dissection using 1% lidocain followed by group I injection of Sodium hyaluronate and group II injection of 40 mg of triamcinolone acetonide, under ultrasound guidance. Baseline VAS pain and nerve conduction study, patient satisfaction, and therapeutic duration, will be determined in 2nd week, 3rd and 6th month after the procedure. US measurements of the median nerve cross-sectional area (CSA) in the CT inlet will be compared pre and post procedure in 6th month and use NCS results as the gold standard diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* patients with mild or moderate carpal tunnel diagnosed by nerve conduction study

Exclusion Criteria:

* secondary carpal tunnel to any other disease and peripheral neuropathy patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
neuropathic pain VAS | 2 weeks
  0-10 VAS scale in the 2nd week after injection

SECONDARY OUTCOMES:
nerve conduction study | 1 month
  motor nerve conduction

OTHER OUTCOMES:
Patient satisfaction | 1month
  (Likert scale) with the grade 1 means that the patient's satisfaction was 30% ,grade 2, the patient's satisfaction was 30-50%,grade 3 ,the satisfaction was 50-80% ,and grade 4 was 80%, Grades 3 and 4 were defined as "overall satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes